CLINICAL TRIAL: NCT00759057
Title: A Clinical Study of the Dynesys(R) Spinal System As a Non-fusion Device for Spinal Stabilization
Brief Title: A Clinical Study of the Dynesys(R) Spinal System
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: PMA not approved. FDA granted permission to close the study.
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: G020291
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Degenerative Spondylolisthesis or Retrolisthesis; Spinal Stenosis; Stenosing Lesion.
Keywords: Spinal Stenosis; Spinal Instability; Leg Pain
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 - Investigational (Experimental): Dynesys Non-Fusion Spinal System
  Interventions: Device: Posterior Pedicle Screw System
- 2 - Control (Active Comparator): Silhouette Posterior Pedicle Screw System as an adjunct to Posterior Lateral Fusion with Autograft.
  Interventions: Device: Posterior Pedicle Screw System

INTERVENTIONS:
Device: Posterior Pedicle Screw System — Implantation of Posterior Pedicle Screw System

SUMMARY:
This non-inferiority study will compare the clinical outcomes of subjects implanted with the Dynesys Spinal System versus the clinical outcomes of subjects implanted with an instrumented posterior lateral spinal fusion.

DETAILED DESCRIPTION:
The purpose of this clinical study is to demonstrate the safety and effectiveness of the Dynesys Spinal System for patients requiring one or contiguous two-level posterior spinal stabilization of the lumbar, and/or sacral spine following decompression. The ability for this implant to maintain spinal alignment and non-fusion of spinal segments, while positively affecting clinical outcomes, will be assessed and compared to a posterior lateral spinal fusion (PLF) procedure using autogenous bone with a semi-rigid, polyaxial posterior spinal fixation system.

ELIGIBILITY:
Inclusion Criteria:

* Patients having degenerative spondylolisthesis or retrolisthesis (up to Grade 1) AND/OR Patients having lateral or central spinal stenosis or other stenosing lesion as diagnosed by radiculopathic signs, neurogenic claudication or imaging studies;
* Candidate for single-level or contiguous two-level PLF between L1-S1;
* Patients have a predominate component of leg rather than back symptoms; symptoms include pain, muscle weakness, and/or sensation abnormality as evidenced by patient history and diagnostic studies.
* Patients may require decompression at the levels considered for treatment
* Pre-operative leg pain score greater than or equal to 40 mm on a 100 mm Visual Analog Scale (VAS);
* Leg pain must be unresponsive to conservative (non-surgical) management for minimum of 3 months;
* Pre-operative Oswestry score greater than or equal to 30 indicating at least moderate disability;
* Skeletally mature individual between ages 20 and 80;
* Must be willing and able to comply with study requirements; including willing and able to sign a study-specific, IRB-approved informed consent form, complete necessary study paperwork and return for required follow-up visits.

Exclusion Criteria:

* Primary diagnosis of discogenic back pain at affected levels as evidenced by a larger back than leg pain component. In the event of multi-level pathology a discogram should be considered;
* Patients with leg pain due to etiologies other than those listed above, such as trauma, peripheral vascular disease and neuropathy should be excluded;
* Degenerative scoliosis greater than 10 degrees at the affected motion segment;
* Supplemental interbody column support (e.g., bone graft, spacers or fusion cages) is planned at the affected level(s);
* Greater than Grade I spondylolisthesis or retrolisthesis at the affected level(s);
* Radiculopathic signs from more than two contiguous or two noncontiguous vertebral body segment(s);
* Previous lumbar fusion attempt(s), previous total facetectomy or trauma at the affected level(s);
* Gross obesity defined as exceeding ideal weight by greater than 40% (measurement details are given in Appendix A);
* Active local or systemic infection;
* Advanced osteoporosis as evidenced by plain film radiographs or history of fractures and confirmed by DEXA scan to confirm adequate bone density;
* Receiving immunosuppressive or long-term steroid therapy;
* Active hepatitis (viral or serum) or HIV positive, renal failure, systemic lupus erythematosus, or any other significant medical conditions which would substantially increase the risk of surgery;
* Documented history of titanium alloy, PET or PCU allergy, or intolerance;
* Active malignancy or other significant medical comorbidities;
* Current chemical dependency or significant emotional and/or psychosocial disturbance that may impact treatment outcome or study participation as evidenced by three or more positive Waddell Signs;
* Pregnancy;
* Incarceration;
* Severe muscular, neural or vascular diseases that endanger the spinal column;
* Missing bone structures, due to severely deformed anatomy or congenital anomalies, which make good anchorage of the implant impossible;
* All concomitant diseases that can jeopardize the functioning and success of the patient;
* Vertebral fractures;
* Treatment of the thoracic and cervical spine;
* Severely deformed anatomy due to congenital anomalies;
* Paralysis

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 399 (Actual)
Dates: Start 2003-03; Primary Completion 2015-06 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Overall Clinical Success (VAS Leg Pain, ODI, Major Complications, Additional Surgical Procedures, Neurological Status) | 24 Months

SECONDARY OUTCOMES:
Radiographic Success, SF-12, Back Pain, Economic and Function Assessment, Subject Perception | 24 Months

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - Scottsdale Spine Center, Scottsdale, Arizona
  - Northwest NeuroSpecialists, Tucson, Arizona
  - Cedars-Sinai Medical Center, The Spine Institute, Los Angeles, California
  - Pacific Regional Neurosurgery, Modesto, California
  - Denver Spine Center, Denver, Colorado
  - Medical Faculty Associates - The George Washington University, Washington D.C., District of Columbia
  - Orthopedic Care & Sports Medicine Center, Aventura, Florida
  - Peachtree Orthopaedic Clinic, Atlanta, Georgia
  - Fort Wayne Orthopedic, Fort Wayne, Indiana
  - Indiana University Neurosurgical, Indianapolis, Indiana
  - Heartland Spine and Hand Center, Overland Park, Kansas
  - Spine Specialty Center (SSC), Baton Rouge, Louisiana
  - Baltimore Neurosurgical Associates, PA, Baltimore, Maryland
  - Orthopaedic Associates, Towson, Maryland
  - Sports Medicine North, Peabody, Massachusetts
  - Orthopedic Consultants, PA, Edina, Minnesota
  - Manhattan Orthopaedics, PC, New York, New York
  - SUNY Upstate Medical University Dept of Orthopedic Surgery, Syracuse, New York
  - Triangle Orthopedic Associates, Durham, North Carolina
  - Orthopaedic Spine Associates, Eugene, Oregon
  - Dept. of Neurosurgery UPMC Presbyterian, Pittsburgh, Pennsylvania
  - Abington Hospital, Willow Grove, Pennsylvania
  - SPINE, Mt. Pleasant, South Carolina
  - College Station Neurosurgery, College Station, Texas
  - Park Plaza Hospital, Houston, Texas
  - SpineMark CRO at TBI, Plano, Texas